CLINICAL TRIAL: NCT01220544
Title: Transplantation of Hematopoetic Stem Cells and Infusion of CD56+CD3- NK Cells From Haploidentical Donors for Patients With Hematological Malignancies
Brief Title: Haploidentical Transplantation With Early Adoptive Transfer of CD56+CD3- NK Cells
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: University of Leipzig (Other)
Responsible Party: Prof. Dr. Lutz Uharek, Charite University Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BELEHAPLO-1412001
Record Dates: First submitted 2010-10-13; First posted 2010-10-14 (Estimated); Last update posted 2010-10-14 (Estimated); Status verified 2010-10

CONDITIONS: Acute Myeloid Leukemias; Advanced Hematological Malignancies; Indication for Allogeneic Stem Cell Transplantation; no HLA-identical Donor Available
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Transplantation, Haploidentical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HaploTransplant with NK cells (Experimental): Haploidentical transplantation of mega-dose CD34+ hematopoetic stem cells with transfer of CD56+CD3-NK cells at day +2
  Interventions: Biological: Haploidentical transplantation with donor NK cells

INTERVENTIONS:
Biological: Haploidentical transplantation with donor NK cells — Pat received a myeloablative conditioning regimen with 12 Gy total-body irradiation in six single doses from day -11 to day -9, thiotepa (5mg/kg/d) on days -8 and -7, fludarabine (40mg/m2/d) from day -6 to day -3, and OKT-3 (5mg/d) from day -5 to day +3. The stem cell graft was aimed to contain > 8 x 10e6 CD34+ cells/kg and < 5 x 10e4 CD3+ cells/kg. A minimum of 1 x 10e7 CD56+CD3- NK cells/kg will be transferred on days +2.

SUMMARY:
Experimental and clinical data suggest that alloreactive NK cells can reduce the risk of graft-rejection, GvHD and leukemic relapse after HLA-mismatched transplantation. The effectiveness of allogeneic NK cells is a function of HLA-differences between donor and recipient that give rise to NK cell clones which do not express inhibitory receptors matching for the HLA molecules of the recipient. Aim of the study is to evaluate cellular therapy with alloreactive, IL-2 activated NK cells after transplantation of T-cell depleted stem cell grafts from one haplotype mismatched family donors in patients with hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML or ALL in first CR with the following high risk features:

  1. AML with aberration Del (5q) -5, del (7q) -7, t(9;22) or t(6;9), abn 3q, 9q, 11q, 20q, 21q, 17p;
  2. AML with a complex caryotype;
  3. secondary AML after previous chemo- or radiotherapy or MDS;
  4. Ph-positive ALL
* Patients with AML or ALL after induction failure or in second CR
* Patients with CML in second chronic or accelerated phase
* Patients with malignant Lymphoma and the following high risk features:

  1. relapse after autologous transplantation
  2. primary chemotherapy refractory disease
* All patients must fulfill the following criteria:

  1. lack of a suitable HLA-identical family, unrelated or cord blood donor
  2. no active infection, no severe impairment of cardial, pulmonary, renal and hepatic function
  3. blast count in the marrow < 30%
  4. informed consent

Exclusion Criteria:

* active infection, no severe impairment of cardial, pulmonary, renal and hepatic function
* blast count in the marrow > 30%
* unable or unwilling to sign and/or understand informed consent

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2001-07; Primary Completion 2010-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate feasibility and safety of alloreactive CD56+/CD3- donor NK cells after one haplotype mismatched transplantation | 1 year
  To evaluate feasibility and safety of cellular immunotherapy with purified alloreactive CD56+/CD3- donor NK cells after one haplotype mismatched hematopoietic stem cell transplantation in patients with high risk hematological malignancies who lack an HLA-identical donor.

SECONDARY OUTCOMES:
transplant related mortality | 1 year
  The investigation of transplant related mortality (incidence of veno occlusive disease; incidence and type of infectious complications).
effectiveness | 2 years
  To evaluate the effectiveness of the therapy (relapse rate; disease free survival; MRD monitoring).
technical aspects of the cell separation procedure | 7 days
  To investigate technical aspects of the cell separation procedure (problems of stem cell mobilization; yield, viability, sterility and purity of the CD34+ and CD56+CD3- cell fraction; log CD3 depletion; in vitro anti-leukemic activity of the CD56+CD3- cell fraction).
stable engraftment of haploidentical stem cell grafts can be achieved after conditioning with total body irradiation, thiotepa, fludarabine and OKT3 and subsequent transfer of megadoses of positively selected CD34+ stem cells and CD56+CD3- NK-cells. | 28 days
  Graft rejection is defined as neutrophils < 0.5 x 10e9/l on day+28 post transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Lutz Uharel, MD, Principal Investigator — Charite University Medicine; Dietger Niederwieser, MD, Principal Investigator — University of Leipzig
Locations (2):
- Germany (2):
  - Charite Campus Benjamin FRanklin, Medical Clinic III, Department of Hematology/Oncology, Berlin, State of Berlin
  - Medical Clinic II, Department of Hematology/Oncology, University of Leipzig, Leipzig